CLINICAL TRIAL: NCT02326597
Title: Comparative Effectiveness of a Decision Aid for Therapeutic Options in Sickle Cell Disease
Brief Title: Decision Aid for Therapeutic Options In Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Lakshmanan Krishnamurti, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00076096a
Record Dates: First submitted 2014-12-18; First posted 2014-12-29 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2017-12

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia; Hemoglobin SS; Hemoglobin SC; Hemoglobin Beta Thalassemia
Keywords: Hydroxyurea; Bone marrow transplant; Chronic blood transfusion; Treatment options for sickle cell disease; Decision making
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin SC Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Practice (Active Comparator): Participants will receive education regarding treatment consideration from their healthcare provider/team as per standard practice (usual care).
  Interventions: Other: Standard Practice
- Standard Practice + Decision Aid (Experimental): Participants will receive standard of care teaching and discussion in addition to web-based decision aid tool access.
  Interventions: Other: Decision Aid Tool; Other: Standard Practice

INTERVENTIONS:
Other: Decision Aid Tool — The tool is a web based decision aid that provides information about the risks and benefits associated with sickle cell disease therapies. Participants will be provided a unique access ID and password to access the information.
  Arms: Standard Practice + Decision Aid
Other: Standard Practice — Standard of care teaching and discussion regarding treatment options given by patient's healthcare provider.

SUMMARY:
Sickle cell disease (SCD) is an inherited disorder with chronic multi-system manifestations affecting 100,000 individuals in the US, largely of minority origin and associated with substantial morbidity, premature mortality, individual suffering, healthcare costs and loss of productivity. Disease modifying treatments such as hydroxyurea, chronic blood transfusion and curative bone marrow transplantation are offered to patients based on physician preference and current practice informed by clinical trials. Decision aids are tools that could help translate evidence from these sources into practice by helping clinicians involve patients in making deliberate choices based on accessible information about the options available and their outcomes and to help them make decisions based on their values and preferences.

The overarching goal of this project is to implement a web based decision aid individualized to patient characteristics to help patients with SCD achieve more accurate perception of risks and benefits of treatment options and make decisions in congruence with their values and preferences. Investigators will use a randomized controlled trial of the effectiveness of a web-based decision aid to give patients accurate information about risks and benefits of therapies that enable patients to make decisions based on their individual values and preferences.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is an inherited disorder with chronic multi-system manifestations affecting 100,000 individuals in the US, largely of minority origin and associated with substantial morbidity, premature mortality, individual suffering, healthcare costs and loss of productivity. Disease modifying treatments such as hydroxyurea, chronic blood transfusion and curative bone marrow transplantation are offered to patients based on physician preference and current practice informed by clinical trials. Decision aids are tools that could help translate evidence from these sources into practice by helping clinicians involve patients in making deliberate choices based on accessible information about the options available and their outcomes and to help them make decisions based on their values and preferences.

There are minimal data about patient-related barriers to and attitudes towards, the use of curative therapies in SCD. Thus significant gaps remain in the understanding of patient perspectives, in the provision of accurate information about risks and benefits of therapies and of incorporating patients' values and preferences in offering treatment options. There is a need for research that helps to understand patient values and preferences and determines how to help patients make informed treatment decision in congruence with their values and preferences.

The overarching goal of this project is to implement a web based decision aid individualized to patient characteristics to help patients with SCD achieve more accurate perception of risks and benefits of treatment options and make decisions in congruence with their values and preferences. Investigators will use a randomized controlled trial of the effectiveness of a web-based decision aid to give patients accurate information about risks and benefits of therapies that enable patients to make decisions based on their individual values and preferences.

Investigators hypothesize that a web based decision aid individualized to patient characteristics can improve knowledge and help patients with SCD achieve more accurate perception of risks and benefits of treatment options and is associated with lower decisional conflict than standard care.

The aims of the study are to estimate the effectiveness of the decision aid tailored to individual patient characteristics on patient knowledge, patient involvement in decision-making and decision-making quality, when compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with sickle cell disease ages 8 to 80 years, inclusive OR
* Parent/legal guardian of patients (age < 18 years) with sickle cell disease who are directly involved in decision making regarding sickle cell disease healthcare treatment OR
* Health care provider directly involved in care of individuals with sickle cell disease, including child of parent/legal guardian enrolled in study
* Patients/parents/caregivers who have made a past decision to not obtain treatment of the considered option or who have not obtained treatment of the chosen option in past 12 months.
* All participants will be able to comprehend English
* Patients/Parent/Legal guardian will have access to the internet from iPad, smart phone or personal computer

Exclusion Criteria:

* Family Members/Individuals/Caregivers not directly involved in decision-making regarding sickle cell disease healthcare.
* Patient/parent/legal guardian who has already made a decision to begin and has started the treatment option.
* Child < 18 years of parent/legal guardian who is participating in Cohort A of this study and randomized to the control arm and not the decision aid arm.
* Spouse, significant other, or other family member involved in decision making for child <18 years if parent/legal guardian of child already enrolled into this study.

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-04-17 (Actual); Study Completion 2017-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmanan Krishnamurti, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Background] Wu CJ, Gladwin M, Tisdale J, Hsieh M, Law T, Biernacki M, Rogers S, Wang X, Walters M, Zahrieh D, Antin JH, Ritz J, Krishnamurti L. Mixed haematopoietic chimerism for sickle cell disease prevents intravascular haemolysis. Br J Haematol. 2007 Nov;139(3):504-7. doi: 10.1111/j.1365-2141.2007.06803.x. No abstract available. PMID 17910640
- [Background] Krishnamurti L, Kharbanda S, Biernacki MA, Zhang W, Baker KS, Wagner JE, Wu CJ. Stable long-term donor engraftment following reduced-intensity hematopoietic cell transplantation for sickle cell disease. Biol Blood Marrow Transplant. 2008 Nov;14(11):1270-8. doi: 10.1016/j.bbmt.2008.08.016. PMID 18940682
- [Background] Rao VK, Price S, Perkins K, Aldridge P, Tretler J, Davis J, Dale JK, Gill F, Hartman KR, Stork LC, Gnarra DJ, Krishnamurti L, Newburger PE, Puck J, Fleisher T. Use of rituximab for refractory cytopenias associated with autoimmune lymphoproliferative syndrome (ALPS). Pediatr Blood Cancer. 2009 Jul;52(7):847-52. doi: 10.1002/pbc.21965. PMID 19214977
- [Background] Aloe A, Krishnamurti L, Kladny B. Testing of collegiate athletes for sickle cell trait: what we, as genetic counselors should know. J Genet Couns. 2011 Aug;20(4):337-40. doi: 10.1007/s10897-011-9366-9. Epub 2011 Apr 19. PMID 21503822
- [Background] Dovey S, Krishnamurti L, Sanfilippo J, Gunawardena S, Mclendon P, Campbell M, Alway S, Efymow B, Gracia C. Oocyte cryopreservation in a patient with sickle cell disease prior to hematopoietic stem cell transplantation: first report. J Assist Reprod Genet. 2012 Mar;29(3):265-9. doi: 10.1007/s10815-011-9698-2. Epub 2012 Jan 5. PMID 22219083
- [Background] Kladny B, Williams A, Gupta A, Gettig EA, Krishnamurti L. Genetic counseling following the detection of hemoglobinopathy trait on the newborn screen is well received, improves knowledge, and relieves anxiety. Genet Med. 2011 Jul;13(7):658-61. doi: 10.1097/GIM.0b013e31821435f7. PMID 21546841
- [Background] Long KA, Thomas SB, Grubs RE, Gettig EA, Krishnamurti L. Attitudes and beliefs of African-Americans toward genetics, genetic testing, and sickle cell disease education and awareness. J Genet Couns. 2011 Dec;20(6):572-92. doi: 10.1007/s10897-011-9388-3. Epub 2011 Jul 12. PMID 21748660
- [Background] Nouraie M, Lee JS, Zhang Y, Kanias T, Zhao X, Xiong Z, Oriss TB, Zeng Q, Kato GJ, Gibbs JS, Hildesheim ME, Sachdev V, Barst RJ, Machado RF, Hassell KL, Little JA, Schraufnagel DE, Krishnamurti L, Novelli E, Girgis RE, Morris CR, Rosenzweig EB, Badesch DB, Lanzkron S, Castro OL, Goldsmith JC, Gordeuk VR, Gladwin MT; Walk-PHASST Investigators and Patients. The relationship between the severity of hemolysis, clinical manifestations and risk of death in 415 patients with sickle cell anemia in the US and Europe. Haematologica. 2013 Mar;98(3):464-72. doi: 10.3324/haematol.2012.068965. Epub 2012 Sep 14. PMID 22983573
- [Derived] Krishnamurti L, Ross D, Sinha C, Leong T, Bakshi N, Mittal N, Veludhandi D, Pham AP, Taneja A, Gupta K, Nwanze J, Matthews AM, Joshi S, Vazquez Olivieri V, Arjunan S, Okonkwo I, Lukombo I, Lane P, Bakshi N, Loewenstein G. Comparative Effectiveness of a Web-Based Patient Decision Aid for Therapeutic Options for Sickle Cell Disease: Randomized Controlled Trial. J Med Internet Res. 2019 Dec 4;21(12):e14462. doi: 10.2196/14462. PMID 31799940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between January 2015 and May 2016.
Pre-assignment Details: Of the 134 participants who signed consent, 120 began study participation and were included in the baseline analysis.
Groups:
- Standard Practice: Participants received education regarding treatment consideration from their healthcare provider/team as per standard practice (usual care).
- Standard Practice + Decision Aid: Participants received standard of care teaching and discussion in addition to web-based decision aid tool access.
Period: Overall Study
Arm/Group | Standard Practice | Standard Practice + Decision Aid
Started | 60 | 60
Completed | 18 | 28
Not Completed | 42 | 32
Not completed — Lost to Follow-up | 42 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Practice | Standard Practice + Decision Aid | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 60 | 120
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 45 | 91
  Male | 14 | 15 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 60 | 60 | 120
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Decision Aid Education Assessed by the Acceptability Survey
Description: Subjects will take an acceptability of education questionnaire which is a 8-item survey to assess the comprehension of education received for the decision aid tool. Each item will be scored on a scale from 1-4 where 1=poor, 2=fair, 3=good, and 4=excellent. Scores will be rated individually 1-4 according to each item. There is no overall total score.
Time Frame: Post Visit 1 (Up to 2 Weeks)
Population: Analysis was completed in both the standard practice and standard practice + decision aid groups together. There were a total of 106 participants who completed the survey.
Measure: Median (Standard Deviation); unit: units on a scale
Groups:
- Standard Practice and Standard Practice + Decision Aid Groups: Participants received standard of care teaching and discussion. Participants received standard of care teaching and discussion in addition to web-based decision aid tool access.
Arm/Group | Standard Practice and Standard Practice + Decision Aid Groups
Number analyzed (Participants) | 106
units on a scale
  Health Impact of Sickle Cell Disease | 3 (.86)
  Risk Factors | 3 (.97)
  Research | 3 (1.1)
  Treatment Options | 3 (1.1)
  Evidence Supporting Self -Care | 3 (1.1)
  Hydroxyurea/BMT/CBT | 3 (1.0)
  Evidence About Hydroxyurea/BMT/CBT | 3 (1.1)
  Stories About Others | 3 (.64)

2. Secondary Outcome: Mean Decisional Self-Efficacy Scale Score
Description: The Decision Self-Efficacy Scale measures self-confidence or belief in one's ability to make decisions, including participate in shared decision making. Items are scored on a scale of 0-4 where 0 is not at all confident and 4 represents very confident.Total scores range from 0 (not at all confident) to 100 (very confident). A score of 0 means 'extremely low self- efficacy' and a score of 100 means 'extremely high self-efficacy.
Time Frame: Month 3, Month 6
Population: Analysis was completed for participants who completed the scale at month 3 and month 6 visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Practice | Standard Practice + Decision Aid
Number analyzed (Participants) | 11 | 16
units on a scale
  Month 3 | 59.29 (22.4) | 75.31 (22.1)
  Month 6 | 71.36 (29.97) | 84.84 (16.39)

3. Secondary Outcome: Mean Difference in Decisional Conflict Scale Scores
Description: Decisional Conflict scale responses are scored for the total score, uncertainty sub-score, informed sub-score, values clarity sub-score, support sub-score and effective decision sub-score. The total score ranges from 0 (no decisional conflict) to 100 (extremely high decisional conflict). The uncertainty sub-score ranges from 0 (feels extremely certain about best choice) to 100 (feels extremely uncertain about best choice). The informed sub-score ranges from 0 (feels extremely informed) to 100 (feels extremely uninformed). The values clarity sub-score ranges from 0 (feels extremely clear about personal values for benefits & risks) to 100 (feels extremely unclear about personal values). The support sub-score ranges from 0 (feels extremely supported in decision making) to 100 (feels extremely unsupported in decision making). The effective decision sub-score ranges from 0 (good decision) to 100 (bad decision).
Time Frame: Baseline, Month 3
Population: Analysis was completed for participants who completed the scale at both baseline and month 3 visits.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Practice | Standard Practice + Decision Aid
Number analyzed (Participants) | 20 | 22
units on a scale
  Total Score | 1.0 [-12.6 to 14.7] | 4.8 [-15.6 to 6.0]
  Uncertainty | .7 [-10.4 to 21.8] | 1.9 [-9.4 to 13.2]
  Informed | -1.3 [-19.2 to 16.5] | -12.1 [-23.3 to -1.0]
  Values Clarity | -.001 [-16 to 16] | -8.0 [-21.4 to 5.5]
  Support | -.4 [-16.3 to 15.4] | 4.6 [-17.7 to 8.6]
  Effective Decision | 1.1 [-10.8 to 13.0] | 2.3 [-14.2 to 9.7]

4. Secondary Outcome: Mean Difference in Decisional Conflict Scale Scores
Description: as for outcome 3
Time Frame: Baseline, Month 6
Population: Analysis was completed for participants who completed the scale at both baseline and month 6 visits.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Practice | Standard Practice + Decision Aid
Number analyzed (Participants) | 16 | 20
units on a scale
  Total Score | 4.6 [-12.0 to 21.1] | -5.0 [-22.4 to 12.4]
  Uncertainty | 7.2 [-10.5 to 25.0] | .8 [-16.2 to 14.6]
  Informed | 1.7 [-18.7 to 22.0] | 10.0 [-32.2 to 12.2]
  Values Clarity | 6.7 [-9.5 to 22.9] | -11.7 [-33.1 to 9.8]
  Support | .6 [-18.2 to 19.4] | 1.3 [-18.1 to 15.6]
  Effective Decision | 6.4 [-11.2 to 24.0] | -2.4 [-19.7 to 14.9]

5. Secondary Outcome: Mean Values Survey Score
Description: The values survey consists of 14 multiple choice questions to measure what is important to a patient when making decisions. The patient decision aid will be tested in the twelve domains of the international patient decision aid standards collaboration criteria checklist. Respondents will be asked to identify perceived importance of individual items (such as procedure related complications, decreasing complication risks, experiencing less pain) and to rate this importance on a 10 point likert scale (0-10) where 1 indicates "not important to me at all" and 10 indicates "extremely important to me". Scores are then converted it to an 11 point scale and averaged.
Time Frame: Post Visit 1 (Up to 2 Weeks)
Population: The analysis includes all participants who completed the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Practice | Standard Practice + Decision Aid
Number analyzed (Participants) | 20 | 22
units on a scale | 10.2 (2) | 10 (1.7)

6. Secondary Outcome: Mean Change in Preparation for Decision Making Scale Score
Description: Preparation for Decision Making Scale assesses a patient's perception of how useful a decision aid or other decision support intervention is in preparing the respondent to communicate with their practitioner at a consultation focused on making a health decision. The preparation for decision-making scale is scored on a 0-100 scale. Higher scores indicate a higher perceived level of preparation for decision making. The total score on the decision making scale is a continuous outcome.
Time Frame: Month 3, Month 6
Population: The analysis includes all participants who completed the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Practice | Standard Practice + Decision Aid
Number analyzed (Participants) | 11 | 16
units on a scale | .48 (.89) | .38 (.74)

7. Secondary Outcome: Mean Knowledge Survey Scores
Description: Knowledge Survey is a 25 multiple choice questionnaire which assesses how much knowledge is being retained after information about risks is received. The knowledge survey is scored as percent correct answers at each time point. This is a set of questions to test knowledge and understanding about sickle cell disease and treatments. As such the answers are dichotomous i.e true or false. The total score of percent correct answers is scored in the range of 0-100%.
Time Frame: Baseline, Month 3, Month 6
Population: The analysis includes all participants who completed the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Practice | Standard Practice + Decision Aid
Number analyzed (Participants) | 38 | 39
units on a scale
  Baseline | 38 (49.87) | 39 (49.83)
  Month 3 | 19 (52.90) | 23 (52.90)
  Month 6 | 46.79 (51.18) | 22 (55.54)

8. Secondary Outcome: Mean Decisional Regret Scale Score
Description: Decision Regret Scale measures distress or remorse after a health care decision. The subject rates regret using a 5 point Likert scale in answering the following questions; 1. It was the right decision 2. I regret the decision 3. I would go for the same decision if I were to do it again 4. The decision caused me a lot of harm 5. It was a wise decision. Total scores range from 0 to 100. A score of 0 means no regret; a score of 100 means high regret.
Time Frame: Visit 3
Population: Number of participants who completed the scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Practice + Decision Aid
Number analyzed (Participants) | 7
units on a scale | 27.5 (23.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study (2 years).
Arm/Group | Standard Practice | Standard Practice + Decision Aid
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT02326597/Prot_SAP_000.pdf